CLINICAL TRIAL: NCT06700837
Title: Impact of Hypoxic Burden on Objective and Subjective Sleepiness in Patients Treated for Obstructive Sleep Apnea
Brief Title: Hypoxic Burden and Sleepiness in Treated OSA Patients
Acronym: MWTBH
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5474
Record Dates: First submitted 2024-09-27; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep; OSA
Keywords: Polysomnography; Polygraphy; Hypoxic burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypoxic burden and Sleepiness in treated OSA patients: In this retrospective study, we reviewed the files of all patients with OSA hospitalised to undergo both polysomnography (PSG) and the 40-min MWT in the Center for Sleep Medicine and Respiratory Disease, Lyon Academic Hospital from September 2017 to January 2020.
  All these patients underwent a full night polysomnography.
  Interventions: Other: Impact of hypoxic burden on objective and subjective sleepiness in patients treated for Obstructive Sleep apnea

INTERVENTIONS:
Other: Impact of hypoxic burden on objective and subjective sleepiness in patients treated for Obstructive Sleep apnea — To determine whether hypoxic load is a predictive marker of objective residual sleepiness measured by MCT in a treated OSAHS population.

SUMMARY:
The Maintenance of Wakefulness Test (MWT) is widely used to objectively assess sleepiness and make safety-related decisions and Epworth Sleepiness Scale (ESS) is the most used scale used to assess subjective sleepiness in sleep medicine.

Besides Obstructive Sleep Apnea measures are rapidly evolving and conventional measures such as apnea-hypopnea index (AHI) and oxygen desaturation index (ODI) are increasingly being supplemented by measures of hypoxia such as hypoxic burden.

Residual AHI in treated OSA have limited predictive value for objective sleepiness. Therefore it seems particularly relevant to identify other predictors of both subjective and objective sleepiness.

This study aims at studying the influence of hypoxic burden as measure of both subjective or objective sleepiness.

We hypothesize that impaired nocturnal oxygenation might influence brain functioning during wakefulness and result in sleepiness as assessed by ESS and MWT.

ELIGIBILITY:
Inclusion Criteria:

* OSA hospitalised to undergo both polysomnography (PSG) and the 40-min MWT in the Center for Sleep Medicine and Respiratory Disease, Lyon Academic Hospital from September 2017 to March 2020.

Exclusion Criteria:

* - age <18 years
* refusal to participate in the study
* diagnosis of central disorder of hypersomnolence
* missing data on the MWT
* Epworth Sleepiness Scale (ESS)
* apnea-hypopnea index (AHI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves consecutive adult patients referred to the Center for Sleep and Respiratory Medicine for performance of MCT from September 2017 to January 2020.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Objective residual sleepiness in a treated OSAHS population as measured by the Multiple Sleep Latency Test (MSLT) in relation to hypoxic load. | 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Pierre TANKERE, MD, Msc, Principal Investigator — Service de médecine du sommeil et des maladies respiratoires Hôpital de la Croix-Rousse
Locations (1):
- Service de médecine du sommeil et des maladies respiratoires Hôpital de la Croix-Rousse, Lyon, France